CLINICAL TRIAL: NCT03588676
Title: Effects of Melatonin on Sleep, Ventilatory Control and Cognition at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert L. Owens (Other)
Responsible Party: Sponsor-Investigator, Robert L. Owens, Associate Physician, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD170200
Record Dates: First submitted 2018-01-03; First posted 2018-07-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Intermittent Hypoxia
Keywords: Hypoxia; High Altitude; Melatonin; Neurocognitive
MeSH Terms: conditions — Hypoxia; Altitude Sickness | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: randomized, placebo controlled, double blind, cross-over trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia (No Intervention): Participants will sleep in room air and receive no melatonin.
- Hypoxia and Placebo (Placebo Comparator): 5mg placebo before sleep study
  Interventions: Other: Placebo
- Hypoxia and Melatonin (Experimental): 5mg melatonin before sleep study
  Interventions: Other: Melatonin

INTERVENTIONS:
Other: Melatonin — 5mg Melatonin
  Arms: Hypoxia and Melatonin
Other: Placebo — 5mg Placebo capsule
  Arms: Hypoxia and Placebo

SUMMARY:
Low oxygen at altitude causes pauses in breathing during sleep, called central sleep apnea. Central sleep apnea causes repeated awakenings and poor sleep. Low oxygen itself and the induced oxidative stress can damage mental function which is likely worsened by poor sleep. Reduced mental function due to low oxygen can pose a serious danger to mountain climbers. However there is also mounting evidence that even in populations of people that live at high altitudes and are considered adapted, low oxygen contributes to reductions in learning and memory. Therefore there is a serious need for treatments which may improve sleep, control of breathing and mental function during low oxygen.Therefore this study aims to determine how melatonin effects control of breathing, sleep and mental performance during exposure to low oxygen.

DETAILED DESCRIPTION:
Research has shown that exposure to low oxygen at altitude causes neurocognitive impairment (impaired mental processing, memory, attention, learning, etc). This impairment in cognitive performance poses a serious risk to mountain climbers and while it has traditionally been thought that people who live at high altitude have adapted to it, evidence shows there is still considerable damage to the brain and impairments in cognitive function of people who live and work at high altitude.

As every cell in the body requires oxygen to survive and function, impairment in cognitive performance at altitude is thought mainly due to reduced oxygen availability to the central nervous system. However, low oxygen at altitude also causes unstable breathing during sleep which results in short periods where the brain stops sending the signal to breath, called central sleep apnea (CSA). During apneas (pauses in breathing) blood oxygen drops even lower and people typically wake up briefly and hyperventilate after apneas. Therefore at altitude people usually get less sleep, their sleep is broken with periods of wakefulness during the night and they experience repeated bouts of severe low blood oxygen levels. Sleep plays a critical role in how the brain repairs and also converts newly acquired information into long-term memory. Therefore broken and reduced sleep can impair cognitive performance, memory and learning. Repeated bouts of severe low oxygen also produces highly reactive molecules that cause damage to cells, called oxidative stress. Oxidative stress also prevents the brain from forming long-term memories and in severe cases (such as extremely high altitude and long duration exposure) can cause neurons in the brain to die. Therefore although sustained low oxygen at altitude likely impairs cognitive function, disturbed sleep and repeated bouts of severely low oxygen likely also contribute to causing brain damage and impaired cognitive performance.

Melatonin is a hormone produced in the pineal gland of the brain during the night which signals to the brain that it is time to sleep. Melatonin is also a very powerful antioxidant which naturally helps to prevent damage in the body from oxidative stress. A study previously reported that melatonin taken 90 mins before bed at 4,300 m (14,200 ft) reduced the time taken to fall asleep, it reduced the number of times people woke up during sleep and improved cognitive performance the following day. However how melatonin caused these effects was not determined. Therefore this study aims to determine how melatonin affects ventilatory control, sleep and neurocognitive performance during sustained hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females
* Age:18-65 years

Exclusion Criteria:

* Sleep Disorders
* Pregnant Females
* Smokers (quit ≥ 1 year ago acceptable)
* Cardiovascular, Pulmonary, Renal, Neurologic, Neuromuscular, or Hepatic Issues
* Diabetes
* Psychiatric disorder, other than mild depression
* Recent exposure to altitude (>8000ft) in the last month or having slept at an altitude >6000ft in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index | 6 weeks
  Measure of Sleep Apnea severity
Neurocognitive Scores | 6 weeks
  Reflex changes between conditions

SECONDARY OUTCOMES:
Loop Gain | 6 weeks
  Measurement of breathing characteristics during sleep using a flow meter attached to a CPAP mask that allows the measurement of expiratory flow
Arousal Threshold | 6 weeks
  requirements for sleep arousal to occur
Sleep Efficiency | 6 weeks
  Time in bed divided by total sleep time
Total Antioxidant Status | 6 weeks
  Measurement taken from blood draw
Hypoxic Ventilatory Response | 6 weeks
  Change in breathing response while breathing low oxygen
Hypercapnic Ventilatory Response | 6 weeks
  Change in breathing response while breathing high carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — Professor; Naomi L Deacon, Ph.D., Study Director — Research Associate; Pamela De Young, Study Chair — Research Associate
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://healthsciences.ucsd.edu/som/medicine/research/centers/sleep-research/research/active-studies/Pages/High-Altitude-and-Sleep.aspx